CLINICAL TRIAL: NCT02321280
Title: Denosumab (A Monoclonal Antibody to Receptor Activator of Nuclear Factor-Kappa B Ligand (RANKL) in Crohn's Disease
Brief Title: The Efficacy of Denosumab in Active Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Toronto (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Charles Bernstein, Distinguished Professor of Medicine, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIC 2014
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm single dose of denosumab (Experimental): Open label = Single dose administration of single dose Denosumab 120 mg subcutaneously
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Single dose subcutaneous administration
  Other Names: Xgeva; Prolia

SUMMARY:
Denosumab, a fully human monoclonal antibody to RANKL was approved for the treatment of postmenopausal osteoporosis in June 2010. It is administered subcutaneously once every 6 months and is highly effective in reducing the risk of vertebral, non-vertebral, and hip fracture risk. There are 3 main concepts underpinning the rationale for using Denosumab to treat CD.

1. CD is associated with an increased risk for osteoporosis and the biology of osteoporosis and T cell mediated inflammation, thought to be integral in CD, involve the RANKL paradigm
2. Animal models of bone loss and colitis treated with RANKL inhibitors improve both bone mass and colitis. A dinitrofluorobenzene sulfonic acid (DNBS) model of colitis in our lab showed significant improvement with Denosumab treatment compared to vehicle (saline) treatment.
3. CD is associated with an increase in mutations at the locus that encodes for RANKL The investigators are conducting an open label pilot study of single dose Denosumab 120 mg s.c. to patients with active Crohn's disease, with assessment of clinical response and remission at 12 weeks.

DETAILED DESCRIPTION:
1.0 Hypothesis Moderate to severely active Crohn's disease (CD) will respond to treatment with Denosumab, (a monoclonal antibody to Receptor Activator of Nuclear factor-Kappa B ligand (RANKL)

The principal research questions to be addressed:

1. Determine if a single dose of Denosumab can induce a clinical response by 12 weeks in persons with active CD 2. Determine if a single dose of Denosumab can induce a clinical remission by 12 weeks in persons with active CD 3. Determine if a single dose of Denosumab can reduce markers of systemic (C-reactive protein, CRP) and intestinal (fecal calprotectin, FCAL) inflammation in persons with active CD.
2. Background Current treatment paradigms of CD involve a step-up approach, where persons with mild disease are treated with 5-aminosalicylate (5-ASA), budesonide or even no therapy. Persons who fail to respond to these relatively inexpensive and well tolerated medications, will often require more intensive therapies including systemic corticosteroids, immunomodulatory agents such as azathioprine or methotrexate, or biologic agents. While the latter have proven efficacy in the treatment of CD, they are quite costly, and their use may result in significant side effects. Currently, the biologic agents infliximab and adalimumab, which specifically antagonize tumor necrosis factor alpha (TNF) are the ultimate step in the medical management of CD. However, nearly one-third of subjects will not respond to a standard anti-TNF based induction regimen, and response can be lost in about one-half of all subjects who responded to the initial induction over the course of one year. Of those who start an anti-TNF and respond, continuous therapy is recommended, the costs of which may exceed $25000-$40000 per year. Furthermore, the combination of an immunomodulator with an anti-TNF agent enhances clinical response, but may increase the risk of infectious complications, and their use is also associated with hepatosplenic T cell lymphoma, which is rare but almost uniformly fatal. In a population based costing study from Manitoba infliximab patients represented a very small proportion of all inflammatory bowel disease (IBD) patients, yet they accounted for a total of approximately $2 million in drug costs in 2005/06, which represented approximately half of all prescription drug costs for IBD patients in Manitoba. Hence, it would be desirable to have a medication that is as effective at inducing and maintaining remission with an improved side effect profile and with a lower cost of provision.

2.1 What is Denosumab: Denosumab, a fully human monoclonal antibody to RANKL was approved for the treatment of postmenopausal osteoporosis in June 2010. It is administered subcutaneously once every 6 months and is highly effective in reducing the risk of vertebral, non-vertebral, and hip fracture risk. A mixed treatment comparison meta-analysis showed Denosumab to be more effective than strontium ranelate, raloxifene, alendronate, and risedronate in preventing new vertebral fractures. It is an agent that works in men as well as women. According to the 2010 Osteoporosis Canada Clinical Practice Guidelines, Denosumab is a first-line option for the pharmacological management of postmenopausal osteoporosis (PMO). "Owing to its efficacy, safety, and potential to improve adherence rates, Denosumab is considered an appropriate first-line pharmacologic option for PMO management." The registration of Denosumab was the culmination of the discovery and clarification of the internal bone microenvironment regulation of bone remodeling: the osteoblast-produced competitors: RANKL and osteoprotegerin (OPG); and the osteoclast receptor: RANK. Our understanding of the pathophysiology of normal bone homeostasis and the pathogenesis of osteoporosis and its integration with the immune response has been greatly advanced by the discovery of RANKL-RANK ligation on osteoblast and osteoclast precursors. Osteoblasts express RANKL which can bind to osteoclast precursors (RANK) or an osteoblast derived soluble decoy receptor -OPG. The binding of RANK to RANKL induces a signaling and gene expression cascade that results in differentiation and maturation of osteoclasts which can ultimately lead to osteoporosis. OPG blocks this interaction, thereby inhibiting osteoclast formation and hence decreases bone resorption. It has been shown that agents that enhance RANKL production are associated with the development of osteoporosis whereas agents that block RANKL reduce bone mineral loss.

When RANKL is upregulated in the estrogen-deficient state and exceeds the amount of OPG, there is an increase in osteoclastogenesis and bone resorption, and this is the major mechanism for bone mass loss and osteoporotic fractures in the postmenopausal state. The human monoclonal antibody to RANKL (Denosumab) was the first product developed to reduce bone resorption by inhibiting RANKL binding to RANK. Denosumab does not accumulate in bone. Extension of the registration trial ('FREEDOM') 5-year data indicates continued safety and efficacy, and this will be extended to 10 years to generate even longer-term data. The profound but reversible suppression of bone turnover that is seen with Denosumab partly explains the continuous increase in bone mineral density seen through 8 years of the phase II clinical trials. As noted above, Denosumab is effective in both men and women and it is potentially effective in glucocorticoid-induced osteoporosis.

2.2 Rationale for Denosumab in CD There are 3 main concepts underpinning the rationale for using Denosumab to treat CD.

1. CD is associated with an increased risk for osteoporosis and the biology of osteoporosis and T cell mediated inflammation, thought to be integral in CD, involve the RANKL paradigm
2. Animal models of bone loss and colitis treated with RANKL inhibitors improve both bone mass and colitis. A dinitrofluorobenzene sulfonic acid model of colitis in our lab showed significant improvement with Denosumab treatment compared to vehicle (saline) treatment.
3. CD is associated with an increase in mutations at the locus that encodes for RANKL

2.2.1 Osteoporosis and IBD: The prevalence of osteoporosis as defined by bone mineral density testing in patients with IBD has been estimated at 15%. Population-based studies show only a modest excess fracture risk in IBD subjects (approximately 20-40% greater than matched controls) and a rate of approximately 1 fracture per 100 patient years. Steroid use is a specific concern in IBD patients-a recent meta-analysis found that current corticosteroid use approximately doubled the risk of fracture independent of risk determined from age and bone mineral density alone. Modulating RANKL in IBD may be effective in managing IBD-associated osteoporosis. RANKL is also a regulator of T cell-dendritic cell interaction in the immune system and is a crucial factor in early lymphocyte development and lymph node organogenesis. The central importance of this system in bone and lymph node homeostasis is seen in RANKL gene-deficient mice which are unable to support osteoclast differentiation, display severe osteopetrosis (even in the presence of bone resorbing factors such as vitamin D3, dexamethasone, and PGE2), show no evidence of bone remodeling, and simultaneously lack all lymph nodes. Activated T cells can directly trigger osteoclastogenesis through RANKL leading to bone loss, an effect that is blocked by OPG. Hence, this system may be critical in linking systemic or mucosal inflammation with altered bone metabolism and, ultimately, osteoporosis.

Denosumab potently removes RANKL from circulation. Denosumab inhibits this pathway by preventing RANKL from binding to its receptor. Denosumab is therefore an antagonist of RANKL's action. Since pharmacologic inhibition of the nuclear factor kappa beta (NF-κB) pathway with infliximab is efficacious for CD, then a repositioning opportunity arises. For safety, cost and compliance reasons Denosumab is an attractive alternative to anti-TNF therapy. The genetic data not only provides additional rationale for the study but focusing on individuals harboring the allele that increases RANKL expression, might provide a cohort that would achieve the greatest gain in being treated with a RANKL inhibitor. Hence we will enroll only patients carrying this G allele, since we hypothesize a slightly larger response to treatment in this subgroup. The risk allele is also relatively common (G-allele frequency = 0.487 in haplotype map (HapMap) CEU), and therefore we expect approximately 75% of patients to be carriers. No clinical trials assessing the effectiveness of Denosumab in the treatment of CD have been undertaken.

2.3 Denosumab safety: Denosumab has been tested in phase III clinical trials in over 10,000 people and has post-marketing surveillance data since 2010. Although nuisance side effects have been reported with denosumab (headache, fatigue, arthralgia), these have not led to clinical sequelae. Hypocalcemia: Anticipated frequency ~2-15% (25-27 ). Reported events of hypocalcemia have been mild, transient and not associated with clinical sequelae. All patients will be recommended to take daily supplemental calcium (≥500mg) and vitamin D (≥400 IU) per day. Serum calcium (corrected for albumin) will be measured 3 days post dose and every 4 weeks. Patients experiencing hypocalcemia will be treated as per the discretion of the treating physician using standard protocols. Osteonecrosis of the Jaw: Anticipated frequency < 1%. The planned dose has been associated with osteonecrosis of the jaw. The concomitant risk factors include cancer, recent or planned invasive dental procedures and current use of anti-angiogenic medications. Individuals with any of these risk factors will be excluded from our trial. Even in trials including only high risk patients (those with cancer), the incidence rates were <2%. All participants will receive written documentation advising them to avoid invasive dental procedures for the duration of the trial, further decreasing the occurrence of this adverse event.

3. The Proposed Trial: An open label multicentred trial. Active therapy arm: Denosumab 120 mg subcutaneously for one dose. This dose of Denosumab has been chosen since it is sufficient to maintain elevated Denosumab levels and depressed RANKL activity as measured by suppression of bone-turnover markers at 3 months post dosing. Further, this dose is the maximal dose clinically used, has a tolerable side-effect profile and adequate pharmacokinetic and pharmacodynamics.

1. CDAI is a calculated score
2. Fecal calprotectin will be measured by ELISA in the lab of the PI.
3. RANKL will be measured by ELISA in the lab of the PI.
4. CRP will be measured as part of routine clinical care in each site's hospital lab.

4. Ileocolonoscopy or abdominal MRI will be undertaken as standard of care in each institution. Each endoscopist will record a CDEIS. Each site will make a disc of each MRI and send to Winnipeg to be read at baseline and study conclusion by a central reader (Dr H Greenberg).

3.6 Sample size: N=30 assuming a 50% response rate has a 95% confidence interval from 33.1 to 66.7%.

3.7 Planned recruitment rate and procedure: Recruitment will occur over a 1 year period. This trial will include 3 Canadian academic sites. We expect to screen 50 subjects and enroll 30 that means screening of 16-18 subjects per site and enrollment of 10 subjects per site. All sites are experienced IBD clinical trial centers and considering the relative ease of the study (single dose) with 16 weeks of follow up we do not anticipate enrollment issues.

Screening Visit: Individuals will be recruited directly from clinical centers specializing in CD care. One gastroenterologist per site will be responsible for clinical care of the patient for the duration of the clinical trial. Clinical study nurses will assess individuals experiencing a CD exacerbation for possible recruitment using a checklist. Potentially eligible patients will have a blood sample drawn and sent to the Innovation Centre (Montreal) for rapid genotyping, which will be completed in 5 business days. If they are carriers of the risk allele, they will undergo an informed consent in person with the study nurse and will then be randomized. Fecal calprotectin and RANKL will be measured centrally at the U of Manitoba.

3.8 Anticipated compliance issues? Since the treatment is a single dose there are no issues with compliance with therapy. In terms of compliance with follow up visits, the visits only require diary review, physical examination and blood draws and occur at 4 weekly intervals after enrollment (except for initial blood draw for serum calcium at day +3).

3.9 Anticipated rate of loss to follow up: We anticipate a loss to follow up of 20% which is a liberal estimate considering the relative ease and duration of the study follow up.

3.10 Proposed type of analyses: Intention to treat. Time to achievement of the primary endpoint will be assessed by Cox proportional hazards and median time to event will be calculated using the Kaplan-Meier method with 95% confidence intervals.

3.11 Proposed frequency of analyses: Single analysis at study conclusion. 3.12 Planned subgroup analyses: We will assess persons with ileal or ileocolonic disease and also separately assess persons with ileocolonic or colonic disease.

3. 13 Follow-up Visits. Serum phosphate, calcium, complete blood count, CRP, electrolytes, fecal calprotectin and RANKL will be measured and all patients will undergo a CDAI. A serum aliquot from each visit will be frozen at -80 degree Celsius for future studies.

3.14 Study Completion Visit: At the 12 week visit, individuals will undergo all assessments done at the 4-weekly visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent.
2. Male or female subjects, 18 to 80 years of age, inclusive.
3. Prior diagnosis of CD confirmed by endoscopy or imaging for > 3 months prior to enrollment with active disease, defined as a Crohn's Disease Activity Index (CDAI) score >220 to <450 and at least one of either: fecal calprotectin >250 ug/g feces, or CRP >8 mg/L.
4. Patients will have evidence of ileocolonic, colonic, or ileal disease that is visualized either endoscopically or on MRI within the prior 6 months.
5. Patients must carry at least one G allele at rs2062305.
6. Patients will be eligible for the study if they are receiving any of the following:

   * mesalamine for >8 weeks with the dose remaining stable for 4 weeks prior to screening;
   * a maximum of 20 mg of prednisone per day (or steroid equivalent), with the dose remaining stable for 2 weeks prior to screening. Steroids must be held stable for the first 4 weeks of the study and then must be tapered by 5 mg per week, to be discontinued entirely by week 8;
   * 6-mercaptopurine, methotrexate or azathioprine for ≥3 months, with the dose remaining stable for 8 weeks prior to screening;

Exclusion Criteria:

1. Monoclonal antibody or experimental agent use within 12 weeks before screening.
2. Use of non-approved drugs for CD.
3. Anticipated need for surgery within 12 weeks
4. Active sepsis, or use of antibiotics within two weeks prior to screening for the treatment of infection.
5. Pregnant, lactating or planning to become pregnant during the study
6. Inability to reliably use birth control for men and women during the course of therapy.
7. Known allergy to Denosumab or ingredients in formulation
8. Treatment of cancer within the last 5 years (except for non-melanoma skin cancers).
9. Recent jaw infection, invasive dental procedures (tooth extraction, dental implants or surgery), anti-angiogenic medications, or hypocalcemia within 1 month prior to screening.
10. Patients will also be excluded if they meet any of the following criteria: Proctocolectomy or total colectomy; stoma; a history of allergy to murine proteins; or treatment with parenteral corticosteroids or corticotropin within four weeks before screening. Serum Hg < 80 g/L, liver enzymes ≥ 2-fold elevated, or other serum biochemistry considered unsafe, or requiring treatment, in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-02; Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Disease Response | week 12
  A drop in CDAI of 100 points

SECONDARY OUTCOMES:
Disease Remission | week 12
  Decrease in CDAI to ≤150 points at 12 weeks.
fecal calprotectin decrease | week 12
  In those with elevated fecal calprotectin at baseline, reduction in fecal calprotectin to <250 ug/g at week 12.
CRP decrease | week 12
  for those with increased CRP at baseline change in CRP to normal at week 12
Endoscopy score decrease | week 12
  For those who underwent endoscopy within 1 month of study enrollment as part of standard of care and who underwent a repeat endoscopy within 1 month of study completion as part of standard of care, improvement in endoscopy by Crohn's Disease Endoscopy Inflammation Score (CDEIS) between baseline and second endoscopy.
MRI improvement | week 12
  For those who underwent abdominal MRI within 1 month of study enrollment as part of standard of care and who underwent a repeat abdominal MRI within 1 month of study completion as part of standard of care then improvement in MRI findings by central reader (Dr H Greenberg) between baseline and second abdominal MRI.
Safety will be assessed for any unforeseen adverse events at each study visit | week 12
  Serum calcium will be assessed at 3 days post drug administration and every 4 weeks. There is a rare incidence of hypocalcemia with use of this drug. Osteonecrosis of the jaw will be assessed at every study visit. This drug is rarely associated with this outcome especially in cancer patients. Liver enzymes every 4 weeks will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Bernstein, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada